CLINICAL TRIAL: NCT00451711
Title: A Randomised, Stratified, Open Label, Phase II Pilot Study on the Safety of a Daily, Intermittent, or Weekly Administration of 1, 3 or 10mg/kg of AmBisome® in Antifungal Primary Prophylaxis of High-Risk Patients With Acute Myeloid Leukaemia
Brief Title: Intermittent Liposomal Amphotericin B Primary Prophylaxis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IN-AU-131-0176
Record Dates: First submitted 2007-03-21; First posted 2007-03-23 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2007-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Prophylaxis; Liposomal Amphotericin B; Acute myeloid leukaemia; Invasive Fungal Infections
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Invasive Fungal Infections | interventions — liposomal amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Liposomal amphotericin B

SUMMARY:
The purpose of this trial is to see which dose of liposomal amphotericin B is the safest when used as a preventer against invasive fungal infection in patients with acute leukaemia who are undergoing chemotherapy.

DETAILED DESCRIPTION:
Invasive Fungal Infections (IFI)are a significant cause of death in patients with acute leukaemia who are undergoing chemotherapy. This is despite improvements in antifungal therapy for the treatment of IFI. The major reason for this is that the current standard diagnostic tests of culture and biopsy lack the ability to make a diagnosis, either early or accurately. Thus other strategies such as the use of prophylaxis are needed. Several antifungal agents have been trialled as prophylaxis but all have disadvantages that limit their effectiveness.

Liposomal amphotericin B(LAB) is a broad spectrum antifungal agent that kills fungal cells. When given in high doses intermittently it supersaturates the liver and the overspill into the bloodstream is absorbed by tissues such as lung, brain and kidneys (i.e. sites where IFI are likely to occur). This effect has been shown in a number of animal and laboratory test-tube studies to reduce fungal burden, improve survival and maintain adequate levels of the drug in between doses. However no intermittent high-dose prophylaxis study has been done in humans. Thus before we proceed to a randomised controlled clinical trial of the efficacy of intermittent high-dose LAB compared with another antifungal agent it is necessary to determine in a phase 2 study which of 2 intermittent dosing LAB regimens (i.e. 3mg/kg three times a week or 10mg/kg once a week) administered during the neutropenic phase of induction-consolidation chemotherapy for treatment of acute leukaemia is safest and best tolerated compared to the standard dosing regimen of 1mg/kg daily of LAB.

Males and females aged >18 years who are undergoing intensive combination chemotherapy for acute leukaemia will be randomised 1:1:1 to either 1mg/kg daily; 3mg/kg 3 times a week or 10mg/kg once weekly of intravenous liposomal amphotericin B. The 3 arms will be compared for the safety of the 3 dosing regimens.

ELIGIBILITY:
Inclusion Criteria:

Patients fulfilling all the following criteria will be eligible:

* Male or female aged >18years;
* Newly diagnosed with acute myeloid leukaemia and undergoing first induction chemotherapy regimen;
* Expected to have absolute neutrophil counts of <0.5x109/L for at least 2 weeks;
* Normal high resolution chest and sinus CT scan at baseline;
* No signs or symptoms of invasive fungal infections
* No prior diagnosis of proven or probable invasive fungal infection within the last 6 months;
* Females of childbearing potential must be: surgically incapable of pregnancy; or practicing an acceptable mode of birth control and have a negative pregnancy test (blood or urine) at baseline;
* Give written informed consent prior to any study-specific procedures;
* Must have the ability and must agree to comply with all study requirements.

Exclusion Criteria:

Patients with any of the following will be ineligible

* Known hypersensitivity to amphotericin B, in particular known history of anaphylactic reaction to amphotericin B;
* Patients undergoing any transplantation;
* Creatinine clearance <60mL/min/1.72 m2;
* Patients with moderate or severe liver disease as defined by aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 5 times the upper limit of normal (ULN)
* Patients who are unlikely to survive more than one month;
* Patients who have received systemic antifungal therapy within the last 15 days
* Any severe cardiovascular disease ( in particular arrhythmias) which may constitute a contra-indication to LAB (AmBisome®) administration;
* Any severe diseases other than acute myeloid leukaemia which in the investigator's judgement may interfere with study evaluations or affect the patients safety;
* Pregnant or nursing females;
* Patients previously included in this study;
* Patients who have taken an investigational drug in the last 30 days prior to the inclusion.
* Patients enrolled in a pre-emptive treatment strategy trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-05; Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Safety as defined by the incidence of all adverse events occurring by the completion of each trial prophylaxis course.

SECONDARY OUTCOMES:
Safety:
Incidence of renal toxicity
Incidence of hepatotoxicity
Incidence of ionic abnormalitities
Incidence of cardiovascular toxicity
Efficacy:
Incidence of proven or probable IFI
Incidence of superficial fungal infections
Incidence of fever of unknown origin requiring empirical antifungal therapy during any course of prophylaxis
Incidence of IFI-related mortality

CONTACTS AND LOCATIONS:
Overall Officials: C. Orla Morrissey, MB, BCh, FRACP, Principal Investigator — The Alfred Hospital, Level 2 Burnet Institute, Commercial Rd., Melbourne, 3004, Victoria, Australia; Anthony P Schwarer, MB, BS, FRACP, MD, FRCPA, Principal Investigator — The Alfred Hospital, Ground Floor South Block, Commercial Rd., Melbourne, Victoria, 3004, Australia
Locations (2):
- Australia (2):
  - The Alfred Hosptial, Melbourne, Victoria
  - Box Hill Hospital, Eastern Health, Melbourne, Victoria